CLINICAL TRIAL: NCT02653911
Title: Efficacy of Acupunture on Menstrual Frequency in Women With Polycystic Ovary Syndrome: Protocol for a Randomized, Controlled Trial
Brief Title: Electroacupuncture on Menstrual Frequency in Women With Polycystic Ovary Syndrome: Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhou Jing, Department of Acupuncture, Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015EC115
Record Dates: First submitted 2016-01-03; First posted 2016-01-13 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Acupuncture
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Bilateral ST25, EX-CA1, CV4 and SP6 will be selected for treatment. After routine sterilization of the local skin, bilateral ST25, EX-CA1, CV4 and SP 6 will be inserted by the needles (0.30 mm in diameter, 40 mm in length) to a depth of 25-30 mm to the abdominal muscle layer with the manipulation of lifting, thrusting and rotating until "de qi". Each session will last for 30 minutes, and the manipulation of lifting, thrusting and rotating evenly three times will be used for CV 4 and SP 6 every 10 minutes. If the date of treatment is during the menstrual circle, the treatment will be continued as usual. Participants will be treated three times a week for 12 weeks with 36 sessions.
  Interventions: Other: Acupuncture
- Sham-acupuncture group (Sham Comparator): The sham ST25, EX-CA1, CV4 and SP 6, which are 1 cun (25 mm) outward to ST25, EX-CA1, CV4 and SP 6, will be inserted to 2-3 mm with needles with a diameter of 0.30 mm and a length of 13 mm. The needles will be inserted without de qi or any manipulation. The treatment sessions will be the same as those in the acupuncture group.
  Interventions: Other: Sham-acupuncture group

INTERVENTIONS:
Other: Acupuncture — Hwato Brand, Suzhou Medical Appliance Factory, China
  Arms: acupuncture group
Other: Sham-acupuncture group — Hwato Brand, Suzhou Medical Appliance Factory, China
  Other Names: Placebo needle
  Arms: Sham-acupuncture group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a dysfunction of endocrine system of women of reproductive age. Approximately 5%-10% women in China have this syndrome. Irregular menstruation (oligomenorrhea or amenorrhea), hirsutism and obesity are the common clinical manifestations of PCOS. The aim of this study is to evaluate the efficacy of acupuncture in improving the menstrual frequency of PCOS patients who do not have fertility requirements.

DETAILED DESCRIPTION:
Methods: A total of 172 participants diagnosed with polycystic ovary syndrome would be randomly assigned to either the acupuncture group or sham-acupuncture group, at a ratio of 1:1. Participants in both groups will receive treatment for 12 weeks, three times a week. The primary outcome will be the proportion of participants with at least a 50% increase from baseline in the monthly menstrual frequency from baseline after 12 weeks intervention, while secondary outcomes will be the difference in anthropometrics, serum hormone level, ovarian morphology, anxiety and depression, and quality of life from baseline to after 12 weeks intervention and to 12 weeks post-intervention follow-up between groups.

Discussion The aim of this study is to evaluate the efficacy and safety of acupuncture for improving menstrual frequency and other symptoms of patients with PCOS. The limitation of this trial is that it would be difficult to blind the acupuncturists. Additionally, these findings may not be suitable for women with PCOS who are seeking pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling any one of the following criteria will be excluded. Participants who fulfill the following criteria will be included.

* Participants meet the Rotterdam diagnostic criteria with oligomenorrhea or amenorrhea. (Oligomenorrhoea is defined as an intermenstrual interval of >35 days or <8 menstrual bleedings in the past year. Amenorrhoea is defined as absent menstrual bleeding or no menstrual bleeding in the previous 90 days.)
* Participants who have at least two of the following features that meet the Rotterdam diagnostic criteria:

  1. Clinical or biochemical hyperandrogenism: Biochemical hyperandrogenaemia is defined as a total serum testosterone concentration above normal threshold, and/or clinical hyperandrogenism is defined as a Ferriman-Gallwey (FG) score of ≥5 or acne defined by the Global Acne Grading System (GAGS) as "mild"/ "moderate"/ "severe"/ "very severe".
  2. Polycystic ovary morphology is defined as the presence of ≥12 follicles in each ovary measuring 2-9 mm in diameter and/or an ovarian volume >10 mL on transvaginal ultrasound.
* Participants who are between 18 to 40 years old.
* Participants who joined the research and provided a signed informed consent voluntarily.

Exclusion Criteria:

* Participants with fertility requirements.
* Participants with oligomenorrhea or amenorrhea caused by hyperandrogenemia, premature ovarian failure, or hypothalamus or pituitary disorders.
* Participants with hyperandrogenism caused by congenital adrenal hyperplasia, Cushing's syndrome and androgen-secreting tumors.
* Participants with endocrine disorders such as thyroid dysfunction, adrenal disorders, hyperprolactinemia and diabetes mellitus.
* Participants with severe heart disease, hepatic disease, renal system and hematopoietic system disease, or malnutrition of the whole body.
* Participants who use hormones or other medications that would affect reproductive function, or received the same protocol of this study in the past three months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who have at least a 50% increase from baseline in monthly menstrual frequency | Months 3
  Baseline monthly menstrual frequency was calculated through the number of menstrual bleeds in three months before intervention divided by three. Monthly menstrual frequency from baseline to three months was calculated through the number of menstrual bleeds during the three month-intervention divided by three.

SECONDARY OUTCOMES:
Change in menstrual frequency | Months 6
  The proportion of participants who have at least a 50% increase from baseline in monthly menstrual frequency
The change in measurements for body mass index (BMI) from baseline | Months 3 and 6
  Change in anthropometry
The change in measurements for waist-hip ratio (WHR) from baseline | Months 3 and 6
  Change in anthropometry
The change in serum luteinizing hormone (LH) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in follicle stimulating hormone (FSH) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in LH/FSH ratio from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in testosterone (T) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in estrogen (E) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in prolactin (PRL) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in progesterone (Prog) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in dehydroepiandrosterone (DHEA) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in sex-hormone binding globulin (SHBG) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in androstenedione (AND) from baseline | Months 3 and 6
  Blood samples will be taken at menstrual cycle days 2-4 when ovulation or bleeding occurs. Otherwise, this will be performed on the arbitrary day of the cycle.
The change in mean difference in ovary volume from baseline | Months 3 and 6
  Change in ovarian morphology
The change in thickness of the endometrium from baseline | Months 3 and 6
  Change in ovarian morphology
The change in the number of follicles <9 mm from baseline | Months 3 and 6
  Change in ovarian morphology
Change in hirsutism | Months 3 and 6
  The change in Ferriman-Gallwey (FG) score from baseline
Change in acne | Months 3 and 6
  The change in Global Acne Grading System (GAGS) from baseline
Change in anxiety and depression | Months 3 and 6
  The change in The score of the Hospital Anxiety and Depression Scale (HADS) from baseline
Change in quality of life | Months 3 and 6
  The change in Polycystic Ovary Syndrome Questionnaire (PCOSQ) scores from baseline

OTHER OUTCOMES:
Blinding assessment | Months 3
  Participants will answer the following questions after 12 weeks of intervention, in order to assess the blinding: "Do you think you have received traditional acupuncture in the past weeks?" The participants can answer "Yes", "No" or "Unclear".
Expectation value of the acupuncture effect assessment | Baseline
  Participants will answer the following questions before the intervention: "Do you think acupuncture will be effective for treating the disease?" "Do you think acupuncture will be effective for improving the related symptoms of PCOS?" The participants can answer "Yes", "No" or "Unclear".
Safety assessment | The whole process
  All adverse reactions will be presented in tables with a description on the categories, severity, rate of incidence, and correlation with the treatment. Adverse reactions related to acupuncture (severe pain, local hematoma, infection and abscess, and retained needle and broken needle during the treatment), including some discomforts after treatment, will be recorded in time in detail. Adverse events irrelevant with the treatment will also be recorded in detail.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Ph D, Study Director — Guang Am Men Hospital,China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No